CLINICAL TRIAL: NCT06118060
Title: The Mechanism of Acupressure on Postoperative Ileus in Patients With Colorectal Cancer Surgery
Brief Title: Acupressure on Postoperative Ileus in Patients With Colorectal Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Yunhong Liu, PhD, Assistant professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KYLL-202307-017
Record Dates: First submitted 2023-10-16; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: acupressure; postoperative ileus
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure group (Experimental): After surgery, the patient is placed in a supine position, exposing both calves, and the operator sits on the edge of the bed and applies acupressure with the thumb or pressing tool (homemade).
  Interventions: Other: Acupressure
- control group (No Intervention): usual care group

INTERVENTIONS:
Other: Acupressure — In this study, the frequency of acupressure was twice a day (the interval between each acupressure was more than 6 hours, 6:00 to 9:00 in the morning and 1:00 to 4:00 in the afternoon); the acupressure was applied from the first day after surgery for a total of 5 days, that is, each patient received a total of 10 acupressure; the duration was 5 minutes, and the bilateral acupressure required 10 minutes.
  Arms: acupressure group

SUMMARY:
The goal of this clinical trial is to learn about acupressure in patients with colorectal cancer surgery. The main questions it aims to answer are:

* whether acupressure can improve the motility of vagus nerve in patients after colorectal cancer surgery
* whether acupressure can reduce the inflammatory response of the body
* whether acupressure can reduce the incidence of gastrointestinal paralysis in patients after colorectal cancer surgery

Participants will receive acupressure at ST36 twice daily starting from the first day after surgery and lasting for five days. Researchers will compare usual care group to see if acupressure has those above effects.

DETAILED DESCRIPTION:
2. Purpose of the study 2.1 Main research objectives: To improve the gastrointestinal function of patients with colorectal cancer after surgery, with the design and implementation of acupressure as the intervention. Through clinical research, the effectiveness of acupressure in improving gastrointestinal function in patients with colorectal cancer surgery will be discussed, and the regulatory effect of acupressure on sympathetic and vagus nerves will be further revealed, and the mechanism affecting gastrointestinal function will be explored from the perspective of nerve and inflammatory response.

2.2 Secondary Research Objectives and Exploratory Research Objectives:

1. To shorten the length of hospital stay, and save medical resources in patients with colorectal cancer surgery;
2. To reveal the mechanism of acupressure, focusing on autonomic regulation and inflammatory response;
3. To explore the association of autonomic regulation with self-reported anxiety, depression, and stress.

3. Study plan 3.1 Design of experiments

1. Investigate the general data and perioperative data of colorectal cancer surgery patients Investigators will independently design the questionnaire, including the following aspects: (1) general information: gender, age, height, weight, previous abdominal surgery history, preoperative radiotherapy and chemotherapy history, underlying diseases, etc.; (2) surgical conditions: surgical method, anesthesia method, duration of surgery, duration of anesthesia, intraoperative heat preservation measures and liquid input, etc.; (3) diet: drinking water, liquid diet, soft diet, ordinary diet time, etc.; (4) exercise: first time out of bed after surgery, etc.; (5) medication: antiemetics, Intramuscular analgesics, etc.
2. Design and implementation of acupressure intervention program On the basis of the previous clinical trial, the technique of acupressure at ST36 will be used to promote gastrointestinal movement compared with control group. The evidence-based basis is mainly derived from domestic and international guideline recommendations, Cochrane systematic review results, meta-analysis results, and large multi-centre randomized controlled trials.
3. Study on the mechanism of acupressure to promote gastrointestinal function By evaluating the 24-hour heart rate variability index of colorectal cancer surgery patients, the regulatory effect of acupressure on autonomic nerve will be evaluated, and the regulatory effect of acupressure on systemic inflammation will be revealed through the changes of postoperative inflammatory factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosis of colorectal cancer;
* Adult patients (age ≥ 18 years);
* Patients undergoing elective surgery, including open surgery, laparoscopic and combined surgery.

Exclusion Criteria:

* Inability to communicate due to language impairment or severe cognitive impairment;
* Skin infection or defect of the lower extremities, which may hinder the localization of ST36 or worsen the infection;
* Plan to perform more than one surgery during hospitalization;
* There are coagulation disorders or peripheral vascular diseases or signs of impaired blood circulation in the lower extremities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | 24 hours after the end of acupressure on day 5
  The differential change of successive heartbeat cycles. Wear a multi-lead Holter (Lepu 12-lead ECG monitor) for 24 consecutive hours.

SECONDARY OUTCOMES:
level of IL-6 | Early morning on the day after the end of acupressure on day 5
  Inflammatory factor. Collect 3 ml of venous blood using a dark green heparin lithium anticoagulant long tube (Item: interleukin 6)
Level of C-reactive protein | Early morning on the day after the end of acupressure on day 5
  Inflammatory factor. Collect 3 ml of venous blood using a purple tube (Item: Blood Cell Analysis Five Classification (Vein) + C-Reactive Protein)
First postoperative exhaust time, defecation time, getting out of bed activity time, drinking time, eating time | Early morning on the day after surgery, up to 5 days
  The time interval between the end of the procedure and the patient's first time of taking these activities.
Bowel motility | Early morning on the day after surgery, up to 5 days
  The outcome assessors will assess the patients' bowel motility on abdominal auscultation by using a stethoscope for one full minute on the body surface above the ileocecal valve in the lower right corner of the abdomen.
Postoperative nausea | Early morning on the day after surgery, up to 5 days
  The outcome assessors will directly asked patients perceived degree of nausea by Numerical Rating Scale (NRS) from 0 to 10 (0 represents no nausea at all and 10 represents the most severe nausea that one can imagine).
Abdominal distension | Early morning on the day after surgery, up to 5 days
  The outcome assessors will directly asked patients perceived degree of abdominal distension by Numerical Rating Scale (NRS) from 0 to 10 (0 represents no bloating at all and 10 represents the most severe bloating that one can imagine).
Abdominal pain | Early morning on the day after surgery, up to 5 days
  The outcome assessors will directly asked patients perceived degree of pain by Numerical Rating Scale (NRS) from 0 to 10 (0 represents no pain at all and 10 represents the most severe pain that one can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Yunhong Liu, PhD, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to yunhongyt@163.com.

REFERENCES:
- [Background] Abodeely A, Schechter S, Klipfel A, Vrees M, Lagares-Garcia J. Does alvimopan enhance return of bowel function in laparoscopic right colectomy? Am Surg. 2011 Nov;77(11):1460-2. PMID 22196657
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Chan HY, Chui YY, Chan CW, Cheng KK, Shiu AT, So WK, Ho SS, Chan MM. Exploring the influence of Traditional Chinese Medicine on self-care among Chinese cancer patients. Eur J Oncol Nurs. 2014 Oct;18(5):445-51. doi: 10.1016/j.ejon.2014.05.005. Epub 2014 Jun 20. PMID 24954767
- [Background] Chao HL, Miao SJ, Liu PF, Lee HH, Chen YM, Yao CT, Chou HL. The beneficial effect of ST-36 (Zusanli) acupressure on postoperative gastrointestinal function in patients with colorectal cancer. Oncol Nurs Forum. 2013 Mar;40(2):E61-8. doi: 10.1188/13.ONF.E61-E68. PMID 23448746
- [Background] Cho S, Shin A, Park SK, Shin HR, Chang SH, Yoo KY. Alcohol Drinking, Cigarette Smoking and Risk of Colorectal Cancer in the Korean Multi-center Cancer Cohort. J Cancer Prev. 2015 Jun;20(2):147-52. doi: 10.15430/JCP.2015.20.2.147. PMID 26151048
- [Background] Drake TM, Ward AE. Pharmacological management to prevent ileus in major abdominal surgery: a systematic review and meta-analysis. J Gastrointest Surg. 2016 Jun;20(6):1253-64. doi: 10.1007/s11605-016-3140-0. Epub 2016 Apr 12. PMID 27073081
- [Background] Fang JY, Dong HL, Sang XJ, Xie B, Wu KS, Du PL, Xu ZX, Jia XY, Lin K. Colorectal Cancer Mortality Characteristics and Predictions in China, 1991-2011. Asian Pac J Cancer Prev. 2015;16(17):7991-5. doi: 10.7314/apjcp.2015.16.17.7991. PMID 26625831
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Martin L, Gillis C, Atkins M, Gillam M, Sheppard C, Buhler S, Hammond CB, Nelson G, Gramlich L. Implementation of an Enhanced Recovery After Surgery Program Can Change Nutrition Care Practice: A Multicenter Experience in Elective Colorectal Surgery. JPEN J Parenter Enteral Nutr. 2019 Feb;43(2):206-219. doi: 10.1002/jpen.1417. Epub 2018 Jul 23. PMID 30035814
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] Wu Z, Boersema GS, Dereci A, Menon AG, Jeekel J, Lange JF. Clinical endpoint, early detection, and differential diagnosis of postoperative ileus: a systematic review of the literature. Eur Surg Res. 2015;54(3-4):127-38. doi: 10.1159/000369529. Epub 2014 Dec 10. PMID 25503902